CLINICAL TRIAL: NCT00678587
Title: Randomised, Double-Blind, Placebo-Controlled, Multi-Centre Study to Evaluate the Safety and Efficacy of Eltrombopag to Reduce the Need for Platelet Transfusion in Thrombocytopenic Subjects With Chronic Liver Disease Undergoing Elective Invasive Procedures
Brief Title: Eltrombopag To Reduce The Need For Platelet Transfusion In Subjects With Chronic Liver Disease And Thrombocytopenia Undergoing Elective Invasive Procedures
Acronym: ELEVATE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: GSK decision
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TPL104054
Record Dates: First submitted 2008-05-13; First posted 2008-05-15 (Estimated); Results first posted 2010-11-08 (Estimated); Last update posted 2018-10-12 (Actual); Status verified 2013-01

CONDITIONS: Non-alcoholic Steatohepatitis; Chronic Liver Disease; HCV; NASH - Nonalcoholic Steatohepatitis; HIV Infection; Thrombocytopenia; Hepatitis C Virus; HBV; Human Immunodeficiency Virus; Liver Diseases; Hepatitis B Virus
Keywords: elective invasive procedure.; platelet transfusion; chronic liver disease-related thrombocytopenia; platelets; thrombopoietin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; HIV Infections; Thrombocytopenia; Hepatitis C; Acquired Immunodeficiency Syndrome; Liver Diseases; Hepatitis B; Jacobs syndrome | interventions — eltrombopag

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo, once daily, oral
  Interventions: Drug: Placebo
- Active (Active Comparator): 75 mg, once daily, oral
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — 75 mg, once daily, oral
  Arms: Active
Drug: Placebo — placebo, once daily, oral
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the ability of eltrombopag to elevate platelet counts thereby reducing the need for platelet transfusions in chronic liver disease patients with thrombocytopenia undergoing elective invasive procedures. The clinical benefit of eltrombopag will be measured by the proportion of subjects who avoid platelet transfusions, before, during and up to 7 days after undergoing an invasive procedure. In addition, bleeding events will be monitored during this time. The number of transfusions, safety events and medical resource utilisation will be monitored during this time and for up to 30 days after undergoing an invasive procedure to help further evaluate clinical benefit.

ELIGIBILITY:
Inclusion Criteria:

* Male and female subjects, 18 years of age or more with chronic liver disease.
* Child-Pugh score of 12 or less.
* Model of End Stage Liver Disease (MELD) score of 24 or less.
* Subjects who, in the opinion of the investigator, are appropriate candidates to undergo an elective invasive procedure and who require a platelet transfusion to manage the risk of bleeding associated with the procedure.
* A baseline platelet count <50,000/µL.
* A baseline serum sodium level >130mEq/L.
* Haemoglobin concentration >8g/dL stable for at least one month.
* A female is eligible to enter and participate in the study if she is of:

Non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:

* Has had a hysterectomy
* Has had a bilateral oophorectomy (ovariectomy)
* Has had a bilateral tubal ligation
* Is post-menopausal (demonstrate total cessation of menses for greater than one year)

Childbearing potential, has a negative urine and/or serum pregnancy test at screening, and within the 24 hour period prior to the first dose of investigational product and uses one of the following acceptable methods of contraception:

* Complete abstinence from intercourse for two weeks before exposure to the study drug, throughout the clinical study, and for 28 days after completion or premature discontinuation from the study to account for the elimination of the study drug (minimum of 5 half-lives).
* Any intrauterine device (IUD) with a documented failure rate of less than 1% per year.
* Double-barrier contraception (condom with spermicidal jelly, or diaphragm with spermicide).
* Male partner who is sterile (diagnosed by a qualified medical professional) prior to the female subject's study entry and is the sole sexual partner for that female.
* Oral contraceptive (either combined or progesterone only).
* Any other contraceptive method with a documented failure rate of <1% per year.
* Subject has no physical limitation to ingest and retain oral medication.
* Subject is able to understand and comply with protocol requirements and instructions and is likely to complete the study as planned.
* Subject is able to provide signed and dated written informed consent.
* In France, a subject will be eligible for inclusion in this study only if either affiliated to or a beneficiary of a social security category.

Exclusion Criteria:

* Subjects with a known hypersensitivity, intolerance or allergy to any of the ingredients in eltrombopag tablets.
* Evidence of portal vein thrombosis on abdominal imaging (ultrasound with Doppler or appropriate MRI/CT imaging techniques) within 3 months of study start.
* History of arterial or venous thrombosis, including Budd-Chiari Syndrome, AND ≥ two of the following risk factors: hereditary thrombophilic disorders (e.g. Factor V Leiden, ATIII deficiency, etc.), hormone replacement therapy, systemic contraception therapy (containing oestrogen), smoking, diabetes, hypercholesterolemia, medication for hypertension or cancer.
* Any disease condition associated with current active WHO Grade 3 or 4 bleeding.
* Active infection requiring systemic antibiotic therapy. Prophylactic use of antibiotics is permitted.
* Pregnant or nursing women.
* Treatment with an investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of study medication.
* History of platelet agglutination abnormality that prevents reliable measurement of platelet counts.
* History of porphyria.
* Previous participation in TPL104054.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2008-06; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (89):
- United States (31):
  - GSK Investigational Site, Birmingham, Alabama
  - GSK Investigational Site, Scottsdale, Arizona
  - GSK Investigational Site, Little Rock, Arkansas
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, San Diego, California
  - GSK Investigational Site, San Francisco, California
  - GSK Investigational Site, Denver, Colorado
  - GSK Investigational Site, Washington D.C., District of Columbia
  - GSK Investigational Site, Jacksonville, Florida
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana
  - GSK Investigational Site, New Orleans, Louisiana
  - GSK Investigational Site, Baltimore, Maryland
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Burlington, Massachusetts
  - GSK Investigational Site, Ann Arbor, Michigan
  - GSK Investigational Site, Detroit, Michigan
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Valhalla, New York
  - GSK Investigational Site, Charlotte, North Carolina
  - GSK Investigational Site, Durham, North Carolina
  - GSK Investigational Site, Portland, Oregon
  - GSK Investigational Site, Hershey, Pennsylvania
  - GSK Investigational Site, Philadelphia, Pennsylvania
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Nashville, Tennessee
  - GSK Investigational Site, Dallas, Texas
  - GSK Investigational Site, Charlottesville, Virginia
  - GSK Investigational Site, Falls Church, Virginia
  - GSK Investigational Site, Richmond, Virginia
- Argentina (5):
  - GSK Investigational Site, Capital Fefderal, Buenos Aires
  - GSK Investigational Site, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - GSK Investigational Site, Derqui, Pilar, Buenos Aires
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
- Belgium (3):
  - GSK Investigational Site, Brussels
  - GSK Investigational Site, Edegem
  - GSK Investigational Site, Ghent
- Canada (4):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Ottawa, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Montreal, Quebec
- France (7):
  - GSK Investigational Site, Clermont Ferrand Cédex 1
  - GSK Investigational Site, Lyon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montpellier
  - GSK Investigational Site, Nice
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Villejuif
- India (2):
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Mumbai
- Italy (11):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, San Giovanni Rotondo (FG), Apulia
  - GSK Investigational Site, Avellino, Campania
  - GSK Investigational Site, Napoli, Campania
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Turin, Piedmont
  - GSK Investigational Site, Palermo, Sicily
  - GSK Investigational Site, Padua, Veneto
- GSK Investigational Site, Lahore, Pakistan
- Poland (5):
  - GSK Investigational Site, Chorzów
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Słupsk
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw
- Russia (4):
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, Samara
  - GSK Investigational Site, Smolensk
  - GSK Investigational Site, Yekaterinburg
- South Korea (3):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Incheon
  - GSK Investigational Site, Seoul
- Spain (9):
  - GSK Investigational Site, Barakaldo
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, L'Hospitalet de Llobregat
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Valencia
  - GSK Investigational Site, Valladolid
- Taiwan (4):
  - GSK Investigational Site, Douliu
  - GSK Investigational Site, Kaohsiung City
  - GSK Investigational Site, Taipei
  - GSK Investigational Site, Taoyuan District

REFERENCES:
- [Derived] Afdhal NH, Giannini EG, Tayyab G, Mohsin A, Lee JW, Andriulli A, Jeffers L, McHutchison J, Chen PJ, Han KH, Campbell F, Hyde D, Brainsky A, Theodore D; ELEVATE Study Group. Eltrombopag before procedures in patients with cirrhosis and thrombocytopenia. N Engl J Med. 2012 Aug 23;367(8):716-24. doi: 10.1056/NEJMoa1110709. PMID 22913681

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Matching placebo
- Eltrombopag 75 mg: Eltrombopag 75 mg administered orally once daily
Period: Overall Study
Arm/Group | Placebo | Eltrombopag 75 mg
Started | 147 | 145
Completed | 127 | 127
Not Completed | 20 | 18
Not completed — Adverse Event | 3 | 3
Not completed — Lack of Efficacy | 1 | 0
Not completed — Protocol Violation | 2 | 1
Not completed — Study Closed/Terminated | 1 | 0
Not completed — Lost to Follow-up | 3 | 5
Not completed — Investigator Discretion | 2 | 6
Not completed — Withdrew Consent | 8 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Eltrombopag 75 mg | Total
Number analyzed (Participants) | 147 | 145 | 292
Age, Continuous [Mean (Standard Deviation); unit: Years] | 53.5 (11.78) | 51.6 (11.04) | 52.5 (11.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 49 | 104
  Male | 92 | 96 | 188
Race/Ethnicity, Customized [Number; unit: participants]
  White | 93 | 85 | 178
  Central/South Asian Heritage | 33 | 41 | 74
  Japanese/East Asian/South East Asian Heritage | 19 | 14 | 33
  African American/African Heritage | 2 | 4 | 6
  Native Hawaiian/Other Pacific Islander and White | 0 | 1 | 1
Number of participants categorized into the indicated Child-Pugh (CP) Class [Number; unit: participants] — The CP score (ranging from 5 to 15; 5=mild, 15=severe), calculated based on total bilirubin, serum albumin, international normalized ratio, ascites, and hepatic encephalopathy, is used to assess liver disease severity. A CP score of 5 or 6 is classified as Class A (mild), a score of 7-9 is classified as Class B (moderate), and a score >=10 is classified as Class C (severe). Participants with a CP score <10 were enrolled in the study. The number of participants analyzed is 140 for placebo and 135 for Eltrombopag; not all participants were compliant and had their baseline CP score measured.
  participants
    Child-Pugh Class A | 59 | 68 | 127
    Child-Pugh Class B | 64 | 57 | 121
    Child-Pugh Class C | 17 | 10 | 27
Model for End-Stage Liver Disease (MELD) Score at Baseline [Median (Full Range); unit: scores on a scale] — MELD uses the following formula to calculate a participant's likelihood of dying within 3 months from liver disease: 3.8 x log (e) (bilirubin milligrams [mg]/deciliter [dL]) + 11.2 x log (e) (international ratio for prothrombin time) + 9.6 log (e) (creatinine mg/dL). Scores range from 6 (least ill) to 40 (most ill): 40 or more, 71.3% mortality; 30-39, 52.6% mortality; 20-29, 19.6% mortality; 10-19, 6.0% mortality; <9, 1.9% mortality. The number of participants analyzed is 140 for placebo and 135 for Eltrombopag; not all participants were compliant and had their baseline MELD score measured.
  scores on a scale | 12 [6 to 25] | 12 [6 to 24] | 12 [6 to 25]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Chronic Liver Disease and Thrombocytopenia (Platelets <50 Gi/L) Who do Not Require a Platelet Transfusion Prior to, During, and up to 7 Days Following Elective Invasive Procedures
Description: A platelet transfusion was given if the platelet count was <50 giga (10^9) per liter (Gi/L) before the procedure. A platelet transfusion was not given if the platelet count was >80 Gi/L (based on a primary endpoint of success). For participants with platelet counts between 50 Gi/L and 80 Gi/L, platelet transfusions were administered at the discretion of the investigator and the physician performing the elective invasive procedure.
Time Frame: Prior to, during, and up to seven days following elective invasive procedures (Study Days 16-19); therefore, this covers a time period from Baseline to Day 26
Population: Intent-to-Treat (ITT) Population: all participants who were randomized to treatment
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 147 | 145
participants | 28 | 104
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 75 mg; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Absolute difference in proportions = 52.8, 95% CI 2-sided [43.2 to 62.4]

2. Secondary Outcome: Number of Participants With a World Health Organization (WHO) Bleeding Score >=2 During and up to 7 Days Following Elective Invasive Procedures
Description: The WHO Bleeding Scale was used to assess bleeding during the study. The range of possible scores is 0 to 4. Grade 0 is no bleeding; Grade 1 is petechiae (small [1-2 millimeter] red or purple spot on the body, caused by a minor hemorrhage); Grade 2 is mild blood loss; Grade 3 is gross blood loss (requiring a transfusion; and Grade 4 is debilitating blood loss (retinal or cerebral associated with fatality).
Time Frame: Prior to, during, and up to 7 days following elective invasive procedures (Study Days 16-19); therefore, this covers a time period from Baseline to Day 26
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 147 | 145
participants | 34 | 25
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 75 mg; Test type: Superiority or Other; Risk Difference (RD) = -5.9, 95% CI 2-sided [-15.1 to 3.3]

3. Secondary Outcome: Number of Participants With the Indicated Number of Platelet Transfusions Administered
Description: Platelet transfusion use was documented at every visit throughout the study from screening until the 4-week (30-day) post-procedure follow-up visit or at the time of participant withdrawal from the study.
Time Frame: Prior to, during, and up to 4 weeks (30 days) following elective invasive procedures (Days 16-19); therefore, this covers a time period from Baseline to Day 26
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 147 | 145
participants
  0 | 30 | 106
  1 | 93 | 24
  2 | 3 | 1
  3 | 2 | 0
  4 | 3 | 0
  5 | 0 | 0
  6 | 1 | 0
  Died/withdrew prior to any platelet transfusions | 15 | 14
Statistical Analysis 1: Comparison: Placebo vs Eltrombopag 75 mg; Test type: Superiority or Other; p < 0.0001, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Median Platelet Count at Screening; Days 1, 8, 15, 16-19; Procedure + 7, 14, 21, 30 Day Follow-up; Early Withdrawal; and Maximum Post-baseline
Description: Procedure +7 = Days 23-26; +14 = Days 30-33; +21 = Days 37-40; +30 = Days 46-49. Early withdrawal can occur at any time. Maximum post-baseline refers to any time point listed above for which the maximum value was reached (therefore this time point is variable).
Time Frame: Screening; Days 1, 8, 15, 16-19; Procedure + 7, 14, 21, 30 day follow-up; early withdrawal; and maximum post-baseline
Population: ITT Population. The number of participants analyzed decreases over time due to missing measurements and to participants dropping out of the study.
Measure: Median (Full Range); unit: Gi/L
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 147 | 145
Gi/L
  Screening, n=147, 145 | 40.0 [8 to 70] | 40.0 [3 to 55]
  Day 1, n=145, 141 | 40.0 [8 to 222] | 40.0 [12 to 62]
  Day 8, n=139, 134 | 41.0 [6 to 190] | 58.5 [20 to 337]
  Day 15, n=132, 131 | 39.0 [6 to 200] | 103.0 [25 to 397]
  Days 16-19, n=50, 49 | 41.5 [18 to 250] | 107.0 [30 to 406]
  Procedure + 7 day follow-up, n=128, 125 | 44.0 [17 to 150] | 148 [30 to 493]
  Procedure + 14 day follow-up, n=116, 125 | 47.5 [13 to 370] | 110 [18 to 805]
  Procedure + 21 day follow-up, n=120, 117 | 44.5 [11 to 200] | 62.0 [15 to 967]
  Procedure + 30 day follow-up, n=125, 127 | 40.0 [10 to 200] | 50.0 [14 to 999]
  Early withdrawal, n=9, 8 | 40.0 [11 to 195] | 41.0 [32 to 140]
  Maximum post-baseline, n=144, 140 | 53.0 [16 to 370] | 152 [32 to 999]

5. Secondary Outcome: Number of Participants With the Indicated Platelet Count at Screening; Days 8 and 15; Procedure + 7, 14, 21, 30 Day Follow-up (FU); and Maximum Post-baseline
Description: as for outcome 4
Time Frame: Screening; Days 8 and 15; Procedure + 7, 14, 21, 30 day follow-up; and maximum post-baseline
Population: as for outcome 4
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 147 | 145
participants
  Screening, <50 Gi/L, n=147, 145 | 133 | 136
  Screening, >=50-<=80 Gi/L, n=147, 145 | 14 | 8
  Screening, >80-<=200 Gi/L, n=147, 145 | 0 | 0
  Screening, >200-<=400 Gi/L, n=147, 145 | 0 | 0
  Screening, >400 Gi/L, n=147, 145 | 0 | 0
  Day 8, <50 Gi/L, n=139, 135 | 98 | 48
  Day 8, >=50-<=80 Gi/L, n=139, 135 | 34 | 50
  Day 8, >80-<=200 Gi/L, n=139, 135 | 7 | 33
  Day 8, >200-<=400 Gi/L, n=139, 135 | 0 | 3
  Day 8, >400 Gi/L, n=139, 135 | 0 | 0
  Day 15, <50 Gi/L, n=132, 131 | 98 | 14
  Day 15, >=50-<=80 Gi/L, n=132, 131 | 26 | 31
  Day 15, >80-<=200 Gi/L, n=132, 131 | 8 | 67
  Day 15, >200-<=400 Gi/L, n=132, 131 | 0 | 19
  Day 15, >400 Gi/L, n=132, 131 | 0 | 0
  Procedure + 7 Day FU, <50 Gi/L, n=128, 126 | 78 | 11
  Procedure + 7 Day FU, >=50-<=80 Gi/L, n=128, 126 | 38 | 20
  Procedure + 7 Day FU, >80-<=200 Gi/L, n=128, 126 | 12 | 60
  Procedure + 7 Day FU, >200-<=400 Gi/L, n=128, 126 | 0 | 30
  Procedure + 7 Day FU, >400 Gi/L, n=128, 126 | 0 | 4
  Procedure + 14 Day FU, <50 Gi/L, n=117, 125 | 63 | 22
  Procedure + 14 Day FU, >=50-<=80 Gi/L, n=117, 125 | 40 | 21
  Procedure + 14 Day FU, >80-<=200 Gi/L, n=117, 125 | 11 | 62
  Procedure + 14 Day FU, >200-<=400 Gi/L, n=117, 125 | 2 | 17
  Procedure + 14 Day FU, >400 Gi/L, n=117, 125 | 0 | 3
  Procedure + 21 Day FU, <50 Gi/L, n=121, 117 | 80 | 38
  Procedure + 21 Day FU, >=50-<=80 Gi/L, n=121, 117 | 30 | 33
  Procedure + 21 Day FU, >80-<=200 Gi/L, n=121, 117 | 10 | 38
  Procedure + 21 Day FU, >200-<=400 Gi/L, n=121, 117 | 0 | 7
  Procedure + 21 Day FU, >400 Gi/L, n=121, 117 | 0 | 1
  Maximum Post-Baseline, <50 Gi/L, n=144, 140 | 60 | 11
  Maximum Post-Baseline, >=50-<=80 Gi/L, n=144, 140 | 53 | 23
  Maximum Post-Baseline, >80-<=200 Gi/L, n=144, 140 | 28 | 62
  Maximum Post-Baseline, >200-<=400 Gi/L, n=144, 140 | 3 | 37
  Maximum Post-Baseline, >400 Gi/L, n=144, 140 | 0 | 7

6. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AEs) and Serious Adverse Event (SAEs) Within the Indicated Category
Description: An AE is any untoward medical occurrence in a patient or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An SAE is any untoward medical occurrence that, at any dose: results in death; is life-threatening; requires hospitalization or prolongation of existing hospitalization; results in disability/incapacity; is a congenital anomaly/birth defect or an ocular event of clinical concern. Medical or scientific judgement is exercised in deciding whether reporting is appropriate in other situations.
Time Frame: Screening to Procedure +30 day follow-up or early withdrawal
Population: Safety population: all randomized participants who received at least one dose of study medication
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 145 | 142
participants
  AEs during study | 85 | 79
  Drug-related AEs in >1 participant | 15 | 31
  Throboembolic AEs | 2 | 6
  Bleeding AEs | 25 | 19
  Hepatobiliary AEs | 16 | 24
  Malignancy AEs | 1 | 1
  Renal AEs | 4 | 2
  Death on study | 2 | 3
  SAEs in >1 participant during study | 17 | 19
  Drug-related SAEs in >1 participant | 4 | 9
  Thrombocytopenia | 1 | 1
  Progression of pre-existing cataract n=145,143 | 2 | 0
  Incident cataract develpment n=145,143 | 2 | 4
  Decrease in visual acuity n=121,124 | 19 | 21
  Renal function abnormality n=145,143 | 27 | 28
  Clinically significant change in ECG n=128,130 | 0 | 1

7. Secondary Outcome: Number of Participants With a Serious Adverse Event That Occurred in Greater Than One Participant
Time Frame: Screening to Procedure +30 day follow-up or early withdrawal
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 145 | 143
participants | 4 | 9

8. Secondary Outcome: Number of Participants With the Indicated Event Relating to Vision
Description: The progression of pre-existing cataracts was measured by the use of slit lamp examination. Decrease in visual acuity is defined as the loss of 3 or more lines of visual acuity in either eye (0.3 log minimal angle of resolution [logMAR], 15 letters on the standard Early Treatment Diabetic Retinopathy Study chart).
Time Frame: Screening or Baseline and at End of Study (Procedure +30 day follow-up or withdrawal visit)
Population: Safety Population: all randomized participants who received at least one dose of study medication. Data are missing for some participants.
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 145 | 143
participants
  Progression of pre-existing cataract, n=145, 143 | 2 | 0
  Cataract development, n=145, 143 | 2 | 4
  Decrease in visual acuity, n=121, 124 | 19 | 21

9. Secondary Outcome: Number of Participants With Renal Function Abnormality
Description: Renal function abnormality was defined by threshold values for: serum creatinine: change from baseline of >=0.3 and <0.5 milligrams (mg)/deciliter (dL) (>=26.6 and <44.3 micromoles [umol]/L) or change from baseline of >=0.5 mg/dL (>=44.3 umol/L); microscopic urine analysis: cellular casts pathologic (as defined by local standards of microscopic urine analysis); urine protein/creatinine ratio (UP/CR): >0.5 mg/mg; Glomerular Filtration Rate (GFR) as determined by the Cockcroft-Gault formula and urine dipstick test.
Time Frame: Screening to Procedure +30 day follow-up or early withdrawal
Population: Safety Population
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 145 | 143
participants | 27 | 28

10. Secondary Outcome: Number of Participants With a Clinically Significant Change in Electrocardiogram (ECG) Results
Description: A 12-lead ECG was obtained in duplicate at screening, baseline, Day 15, and withdrawal from the study. Participants rested supine for 5 minutes before the 12-lead ECG was recorded. A 30 second rhythm strip was obtained, and the ECG was calibrated, labelled, and initialled by the person performing the recording. A written, interpretive assessment detailing clinical significance was produced, dated, and signed off by the physician at the site.
Time Frame: Screening, Baseline, Day 15, and Withdrawal
Population: Safety Population. Data were missing for some participants.
Measure: Number; unit: participants
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 128 | 130
participants | 0 | 1

11. Secondary Outcome: Pharmacokinetics (PK) of Eltrombopag, Steady State AUC(0-tau)
Description: AUC(0-tau) is the area under a concentration versus time curve between dose interval following repeat dosing. It is a measure of systemic drug exposure.
Time Frame: Day 14
Population: PK Subpopulation: all participants who were treated with eltrombopag and provided evaluable PK samples
Measure: Geometric Mean (95% Confidence Interval); unit: hour*micrograms (ug)/milliliter (mL)
Arm/Group | Eltrombopag 75 mg
Number analyzed (Participants) | 41
hour*micrograms (ug)/milliliter (mL) | 250 [211 to 296]

12. Secondary Outcome: Pharmacokinetics (PK) of Eltrombopag, Cmax
Description: Cmax is the steady state peak plasma concentration of a drug observed after its administration.
Time Frame: Day 14
Population: PK Subpopulation
Measure: Geometric Mean (95% Confidence Interval); unit: ug/mL
Arm/Group | Eltrombopag 75 mg
Number analyzed (Participants) | 41
ug/mL | 11.6 [9.8 to 13.6]

13. Secondary Outcome: Pharmacokinetics (PK) of Eltrombopag, t1/2
Description: t1/2 is the half life of a drug based on its terminal phase. Half life is defined as the time necessary to halve the plasma concentration.
Time Frame: Day 14
Population: PK Subpopulation
Measure: Geometric Mean (95% Confidence Interval); unit: hours
Arm/Group | Eltrombopag 75 mg
Number analyzed (Participants) | 41
hours | 70.3 [60.7 to 81.5]

14. Secondary Outcome: Pharmacokinetics (PK) of Eltrombopag, CL/F
Description: CL/F is the apparent plasma clearance, where CL is an estimate of the total body clearance, and F is the fraction of dose absorbed. Total clearance is the volume of blood cleared of the drug by the various elimination processes (metabolism and excretion) per unit time.
Time Frame: Day 14
Population: PK Subpopulation
Measure: Geometric Mean (95% Confidence Interval); unit: Liters/hour
Arm/Group | Eltrombopag 75 mg
Number analyzed (Participants) | 41
Liters/hour | 0.30 [0.25 to 0.36]

15. Secondary Outcome: Mean Number of Days Spent in the Hospital
Description: The number of days spent in the hospital was analyzed as an indication of medical resource utilization throughout the study.
Time Frame: as for outcome 3
Population: ITT Population. Data are missing for some participants.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 144 | 144
days | 1.3 (3.77) | 1.7 (6.43)

16. Secondary Outcome: Mean Number of Unscheduled Office Visits, Unscheduled Laboratory Tests, and Unscheduled Procedures
Description: The number of unscheduled events was analyzed as an indication of medical resource utilization throughout the study.
Time Frame: as for outcome 3
Population: ITT Population. Data are missing for some participants.
Measure: Mean (Standard Deviation); unit: unscheduled events
Arm/Group | Placebo | Eltrombopag 75 mg
Number analyzed (Participants) | 144 | 144
unscheduled events
  Unscheduled office visits | 0.8 (1.64) | 1.0 (2.91)
  Unscheduled laboratory tests | 1.1 (3.78) | 1.8 (5.67)
  Unscheduled procedures | 0.3 (0.81) | 0.4 (1.65)

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) with an onset on or after the start date of study medication were collected until the end of the study (up to the end of Week 7).
Description: The Safety Population, comprised of all randomized participants who received at least one dose of study medication, was used for the collection of AEs and SAEs.
Arm/Group | Placebo | Eltrombopag 75 mg
Serious Adverse Events (participants affected / at risk) | 17/145 | 19/143
Other Adverse Events (participants affected / at risk) | 35/145 | 40/143
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Eltrombopag 75 mg (N=143)
Mesenteric vein thrombosis (Gastrointestinal disorders) | 1 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Appendix disorder (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Ileus paralytic (Gastrointestinal disorders) | 0 | 1
Colitis ischaemia (Gastrointestinal disorders) | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Oesophageal haemorrhage (Gastrointestinal disorders) | 0 | 1
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Peritonitis (Gastrointestinal disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 2 | 0
Cataract (Eye disorders) | 3 | 1
Macular degeneration (Eye disorders) | 0 | 1
Visual accuity reduced (Eye disorders) | 0 | 1
Sepsis (Infections and infestations) | 0 | 2
Appendicitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1
Gastroenteristis (Infections and infestations) | 1 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 1
Peritonitis acute (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 3 | 2
Encephalopathy (Nervous system disorders) | 1 | 1
Portal vein thrombosis (Hepatobiliary disorders) | 2 | 4
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hepatic hydrothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Thrombocytosis (Blood and lymphatic system disorders) | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 1
Acute myocardial infaction (Cardiac disorders) | 1 | 0
Pyrexia (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Shock (Vascular disorders) | 1 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0
Fluid retention (Metabolism and nutrition disorders) | 0 | 1
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=145) | Eltrombopag 75 mg (N=143)
Headache (Nervous system disorders) | 6 | 11
Pyrexia (General disorders) | 10 | 8
Abdominal pain (Gastrointestinal disorders) | 7 | 7
Nausea (Gastrointestinal disorders) | 7 | 7
Diarrhoea (Gastrointestinal disorders) | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.